CLINICAL TRIAL: NCT05699096
Title: Perfluorooctyl Bromideessential for Repositioning Giant Retinal Breaks and Can be Used for Removal of Subretinal Fluid as Well as Stabilization of the Retina to Offset
Brief Title: Perfluorooctyl Bromide Which Empowers the Liquid to Flat the Detached Retina and Displace the Underneath Fluids Anteriorly
Status: Recruiting | Type: Observational
Sponsor: EL Romany Ophthalmics Factory (Industry)
Responsible Party: Sponsor
Other Study IDs: ROPFO
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- eye surgery ,Vitreoretinal Surgery and Related Ocular Inflammation

SUMMARY:
Perfluorohexyloctaneis Essential for Repositioning Giant Retinal Breaks and Can be Used for Removal of Subretinal Fluid as Well as Stabilization of the Retina to Offset

ELIGIBILITY:
Inclusion Criteria:

* - Is 20 years or older Has been diagnosed with Keratoconus; Has no other active ocular disease; Is not pregnant or nursing;

Exclusion Criteria:

* Is under the age of 20 Has best corrected visual acuity outside 20/400; Pregnant or nursing at the time of enrollment in the study;

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
flat the detached retina and displace the underneath fluids anteriorly | Base line
  the effect of Perfluorooctyl Bromide on the retina ,under ophthalmic microscope check the flatted retina

CONTACTS AND LOCATIONS:
Locations (1):
- Girgis Boules, Cairo, Kubri EL Kubba, Egypt